CLINICAL TRIAL: NCT06447753
Title: COMPARATIVE EVALUATION OF DIRECT PULP CAPPING AND COMPLETE PULPOTOMY IN MATURE PERMANENT MANDIBULAR MOLARS WITH CLINICAL SIGNS INDICATIVE OF MODERATE PULPITIS: RANDOMIZED CLINICAL TRIAL
Brief Title: COMPARATIVE EVALUATION OF DIRECT PULP CAPPING AND COMPLETE PULPOTOMY IN MATURE PERMANENT MANDIBULAR MOLARS WITH CLINICAL SIGNS INDICATIVE OF MODERATE PULPITIS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Sakshi
Record Dates: First submitted 2024-06-02; First posted 2024-06-07 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Moderate Pulpitis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Direct pulp capping (Experimental)
  Interventions: Procedure: Direct pulp capping
- Complete pulpotomy (Active Comparator)
  Interventions: Procedure: Complete Pulpotomy

INTERVENTIONS:
Procedure: Direct pulp capping — after caries excavation, the pulp will be inspected visually. If bleeding present, sterile cotton soaked in 3% NaOCl will be placed over the pulpal wound for 2 minutes, repeated for up to 6 min if required. Cases in which bleeding will not stop within 6 minutes will be excluded from the study and further managed by RCT. The exposed pulp will be capped with MTA which will be freshly mixed according to manufacturer's instructions and placed in thickness of 2 to 3 mm over the pulp exposure site using an amalgam carrier following which the cavity floor will be dabbed with moist sterile cotton pellet to ensure the setting of MTA, followed by application of a layer of light-cure RMGIC over MTA and light-curing for 20s. Then tooth will be restored using composite resin following etch and rinse technique.
  Arms: Direct pulp capping
Procedure: Complete Pulpotomy — exposed pulp tissue will be amputated using fresh sterile large round diamond bur in a high-speed hand-piece under water coolant 28to the level of canal orifices. The pulp wound will be irrigated with 3% NaOCl. For hemostasis, sterile cotton soaked in 3% NaOCl will be placed over the pulpal wound for 2 minutes, repeated for up to 6 min if required. Root canal therapy will be initiated in cases in which haemostasis is not achieved within 6 minutes. After hemostasis, ProRoot MTA will be placed in thickness of 2 to 3 mm over the pulp exposure site using an amalgam carrier. After placement, the cavity floor will be dabbed with moist sterile cotton pellet to ensure the setting of MTA, followed by application of a layer of light-cure RMGIC over MTA and light-curing for 20s. The tooth then will be restored using composite resin following etch and rinse technique.
  Arms: Complete pulpotomy

SUMMARY:
Title: Comparative evaluation of direct pulp capping and complete pulpotomy in mature permanent mandibular molars with clinical signs indicative of moderate pulpitis: Randomized Clinical Trial

Rationale: According to new Wolters pulpal clinical classification, Moderate pulpitis exhibit symptoms of prolonged reaction to cold, which can last for minutes, possibly percussion sensitive and spontaneous dull pain which are correspond to irreversible pulpitis.

Complete/partial pulpotomy are suggested to be the choice of treatment for such cases. It has been suggested that infection is often the cause of inflammation, an inflamed pulp should be able to heal if the source of infection is eliminated as in other body organs. Removal of trigger (i.e. caries) followed by application of biocompatible material which makes a good seal in a sterile environment has potential to allow for recovery and healing of the inflamed pulp tissue which is thought to be beyond recovery. Based on this premise, DPC can be considered as minimally invasive approach for the management of teeth with inflamed pulps in place of the conventional approach of partial/complete pulpotomy in adults

Research Question Does Direct Pulp Capping have comparable outcome with complete pulpotomy in mature permanent teeth with clinical signs indicative of moderate pulpitis?

DETAILED DESCRIPTION:
Rationale: Vital pulp therapy has been traditionally recommended only in teeth with reversible pulpitis with no periapical pathologies or in teeth with either mechanical pulp exposure or recent traumatic exposure. Clinical symptoms such as characteristic, severity and intensity of pre-operative pain do not accurately talk about the status of the pulp inflammation and the depth of involvement. It has been demonstrated that there is no precise correlation between clinical symptoms and the histopathological status of the pulp, mainly in case of irreversible pulpitis, that might lead to a wrong diagnosis. Vitality tests such as cold test or electric pulp tests reveal only whether the pulp is responsive to respective stimuli or not. According to new Wolters pulpal clinical classification, Moderate pulpitis exhibit symptoms of prolonged reaction to cold, which can last for minutes, possibly percussion sensitive and spontaneous dull pain which are correspond to irreversible pulpitis.

Complete/partial pulpotomy are suggested to be the choice of treatment for such cases. It has been suggested that infection is often the cause of inflammation, an inflamed pulp should be able to heal if the source of infection is eliminated as in other body organs. Removal of trigger (i.e. caries) followed by application of biocompatible material which makes a good seal in a sterile environment has potential to allow for recovery and healing of the inflamed pulp tissue which is thought to be beyond recovery. Based on this premise, DPC can be considered as minimally invasive approach for the management of teeth with inflamed pulps in place of the conventional approach of partial/complete pulpotomy in adults

Aim: To compare the outcome of direct pulp capping and complete pulpotomy in mature mandibular permanent molars with clinical signs indicative of moderate pulpitis.

Objectives:

1. To evaluate the clinical and radiographic success of direct pulp capping in mature permanent molars with clinical signs indicative of moderate pulpitis.
2. To evaluate the clinical and radiographic success of complete pulpotomy in mature permanent molars with clinical signs indicative of moderate pulpitis.
3. To evaluate pain incidence and severity after direct pulp capping and complete pulpotomy in mature permanent molars with clinical signs indicative of moderate pulpitis

P (Population) - Mature Permanent Mandibular molars with clinical signs of moderate pulpitis I (Intervention) -Direct pulp capping C (Comparison) - Complete pulpotomy O (Outcome) - Assessment of clinical and radiographic success at 12 months follow up.

* To assess incidence and reduction in pain post operatively at every 24 hours till 1 week

ELIGIBILITY:
Inclusion Criteria:

1. The patient should be ≥18 years of age. 2. Restorable mature permanent 1 st and 2nd Mandibular molars with extremely deep caries (≥2/3 dentine involvement) 3. Tooth should give positive response to pulp sensibility testing. 4. Clinical diagnosis of moderate pulpitis. 5. Radiographic finding of periapical index (PAI) score ≤2. 6. Healthy periodontium (probing pocket depth ≤3 mm and mobility within normal limit).

-

Exclusion Criteria:

1. Teeth with immature roots.
2. No pulp exposure after caries excavation.
3. Bleeding could not be controlled in 6 minutes.
4. Signs of pulpal necrosis, sinus tract, swelling, insufficient bleeding after pulp exposure.
5. History of analgesic intake in previous 1 week, or antibiotic intake in 1 month.
6. Internal/external resorption.
7. Contributory medical history (alcoholism, smokers, diabetic, hypertension, drug dependency, Heart or valve disease, hepatitis, herpes, immunodeficiency (HIV), infectious diseases, kidney or liver, migraine) -

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 92 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Clinical and radiographic success | 12 months
  Clinical success criteria No history of spontaneous pain or discomfort except for the initial days after treatment.
  No tenderness to palpation or percussion and the tooth is functional. Normal mobility and probing pocket depth. Soft tissues around tooth are normal with no swelling or sinus tract. Radiographic success criteria No pathosis evident on the radiograph such as root resorption, furcal pathosis or new periapical pathosis. Periapical Index score 1 or 2 according to Orstavic6 et al.

SECONDARY OUTCOMES:
Pain incidence and reduction | 7 days
  Patients will be informed that they may experience pain in the days after treatment and will be instructed to record their pain at 24 h, 2, 3, 4, 5, 6 and 7 days after the treatment, to be submitted after 1 week. They will be instructed to use analgesics (Ibuprofen 400 mg every 6-8 h), if needed for pain relief. They will be requested to note down the details of analgesic intake on the pain form regarding the number of doses required, timing of the dose and whether it provided adequate pain relief or not (yes/no). 29 Visual analogue scale (VAS) from 0 to 100 will be used to record preoperative and post
  -operative pain.

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay Tewari, MDS, Study Director — pgids rohtak
Locations (1):
- PGIDS, Rohtak, Haryana, India